CLINICAL TRIAL: NCT01129830
Title: The Effect of DHEA on Markers of Ovarian Reserve in Women With Diminished Ovarian Reserve
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Suboptimal recruitment
Sponsor: Virginia Center for Reproductive Medicine (Other)
Responsible Party: Principal Investigator, Fady I. Sharara, M.D, Medical Director, Virginia Center for Reproductive Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VCRM 3
Record Dates: First submitted 2010-05-19; First posted 2010-05-25 (Estimated); Last update posted 2014-09-22 (Estimated); Status verified 2014-09

CONDITIONS: Infertility
Keywords: ovarian reserve; FSH; anti-mullerian hormone; estradiol; oocyte; IVF; embryo transfer
MeSH Terms: conditions — Infertility | interventions — Dehydroepiandrosterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dehydroepiandrosterone (Other): infertile women with low anti mullerian hormone levels
  Interventions: Dietary Supplement: dehydroepiandrosterone

INTERVENTIONS:
Dietary Supplement: dehydroepiandrosterone — DHEA supplementation 25 mg tid for 3 months

SUMMARY:
This prospective study evaluates the effect of DHEA supplementation on markers of ovarian reserve in women with diminished ovarian reserve.

DETAILED DESCRIPTION:
Ovarian reserve markers, such as FSH, estradiol, AMH, ovarian volume and antral follicle counts will be monitored on DHEA supplementation in a prospective fashion.

ELIGIBILITY:
Inclusion Criteria:

* infertile women with diminished ovarian reserve

Exclusion Criteria:

* women > 45

Ages: 21 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2010-01; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
live birth rate | 3 years
  Live birth rate will be monitored for women who took DHEA supplementation

SECONDARY OUTCOMES:
number of oocytes | 3 years
  Number of retrieved oocytes for patients undergoing IVF will be monitored along with ovarian response

CONTACTS AND LOCATIONS:
Overall Officials: Fady I Sharara, M.D, Principal Investigator — Virginia Center for Reproductive Medicine
Locations (1):
- Virginia Center for Reproductive Medicine, Reston, Virginia, United States

REFERENCES:
- [Background] Barad D, Brill H, Gleicher N. Update on the use of dehydroepiandrosterone supplementation among women with diminished ovarian function. J Assist Reprod Genet. 2007 Dec;24(12):629-34. doi: 10.1007/s10815-007-9178-x. Epub 2007 Dec 11. PMID 18071895